CLINICAL TRIAL: NCT04794309
Title: Effect of Circuit Training With Low-carbohydrate Diet on Body Composition, Cardiometabolic Indices, and Exercise Capacity in Young Males With Mild to Moderate Obesity in Saudi Arabia
Brief Title: Outcomes of Circuit Training and Low Carbohydrates Diet in the Young Obese Male in KSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Lecturer, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUREC-Apr.11/COM-2017/15
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: Seventy young males with obesity participated in this study. They were divided randomly into two groups. Group 1 received circuit training with low-carbohydrate (LC) diet intervention and Group 2 was the control group. The study variables such as exercise capacity, body composition, skinfold thickness, percentage of body fat (BF%), and lipid profile were measured at the baseline and at the end of a 12-week intervention.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The participants will receive circuit training exercise and dietary intervention.
  Interventions: Other: Circuit training exercise; Dietary Supplement: Healthy high Fiber diet
- Control group (Active Comparator): The participants will be only involved in dietary intervention.
  Interventions: Dietary Supplement: Healthy high Fiber diet

INTERVENTIONS:
Other: Circuit training exercise — circuit training exercise start with 5 minutes of warming-up then followed by a 30-minute conditioning protocol formed 20 minutes of aerobic exercise and 10 minutes of resisted exercise. The cool-down period is doing in form of walking on a treadmill in low intensity for 5 minutes.
  Aerobic exercise will be performed on an electronically-braked cycle ergometer (Quinton Excalibur, QuintonInstrument Company, Bothell, WA). resistance exercise (RT) in the form of eight different exercises will be performed during each workout: military press, leg extension, bench press, standing leg curl (ankle weights), lateral pull-down, dumbbell triceps push-down, dumbbell seated biceps curl, and sit-ups (abdominal curls).
  The participant will do 10 minutes for Aerobic exercise followed by 10 minutes of resistance exercise then 10 minutes for Aerobic exercise. This cycle training will perform five days per week for eight weeks.
  Arms: Experimental Group
Dietary Supplement: Healthy high Fiber diet — The diet will be tailor-made for the individual for the body type and obesity in consultation with the nutritionist.

SUMMARY:
Obesity is one of the common public problems that its prevalence increase incredibly in the last three decades in KSA. Thirty obese males aged 20 to 39 years will participate in the study. The participants will be evaluated on skinfold thickness, percent of body fat, lipid profile, and exercise capacity. All participants will perform a circuit training of aerobic and resistance exercises and be instructed to follow a low carbohydrate diet for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Obese young male subjects with a mass index between BMI >30 kg/m2 and 40 kg/m2).
2. Subjects ages range from 20 to 39 years.
3. Previously sedentary, defined as no strength training and less than 150 minutes of brisk walking or moderate exercise per week and < less than 60 minutes of vigorous exercise per week in the preceding 6 months.
4. Only subjects who are nonsmokers.
5. Subjects who are not taking insulin.
6. Had no evidence or history of coronary artery disease.

Exclusion Criteria:

1. Subjects were excluded if they reported a history of heart disease, respiratory conditions, stroke, diabetes, recent cancer, other life-threatening illness, or any condition that limited their ability to engage in moderate-intensity exercise.
2. Smoking

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic index | 12 weeks
  High-density lipoprotein, low-density lipoprotein, triglycerides, and total cholesterol will be evaluated through a blood sample from the participants at the start and at the end of 12 weeks of intervention.
Exercise capacity | 12 weeks
  The renowned modified sub-maximal treadmill exercise test,which is the leading indicator of EC,was done to calculate maximum oxygen uptake (VO2max). The test began with a warm-up at a speed of 2.7 km/h for five minutes, andthe speed was increasedevery three minutes until the participantexerted the maximum effort and stopped upon exhaustion.
Body Weight | 12 weeks
  Measured in kilograms
Height | 12 weeks
  Measured in meters
Body mass index | 12 weeks
  Measured in kg/m^2
Waist circumference | 12 weeks
  Measured in centimeters
Hip circumference | 12 weeks
  Measured in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Majmaah University, Majmaah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The Data will be available when the article gets published in a journal.